CLINICAL TRIAL: NCT02813668
Title: Worksite Lifestyle Program for Reducing Diabetes and Cardiovascular Risk in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Public Health Foundation of India (Other); Madras Diabetes Research Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mary Beth Weber, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00080327; R01HL125442 (NIH)
Record Dates: First submitted 2016-06-17; First posted 2016-06-27 (Estimated); Results first posted 2023-09-08 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Diabetes; Heart Disease; Obesity
Keywords: Nutrition; Occupational Health
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle Intervention Training Program (Experimental): Participants at risk for developing diabetes or with unmedicated diabetes will participate in a lifestyle intervention training program. Individuals in the training program, as well as un-enrolled workers at the study sites, will be exposed to positive changes at the worksite to promote increased physical activity and healthier diets.
  Interventions: Behavioral: Lifestyle Intervention Training Program

INTERVENTIONS:
Behavioral: Lifestyle Intervention Training Program — Participants will be placed into a peer-led classes of 10 to 12 people. The curriculum contains sixteen core sessions that occur weekly for four months followed by an eight month maintenance period. During lifestyle classes, participants will learn strategies for eating a healthy diet, increasing physical activity, overcoming barriers, building social support, reaching and maintaining a healthy wait, and maintaining healthy blood glucose levels. Participants will also be assigned goals to achieve; increasing physical activity and losing 5% of their baseline body weight. During maintenance, participants will receive biweekly SMS text messages providing lifestyle advice tips and encouragement.

SUMMARY:
This study will test the implementation, effectiveness, cost-effectiveness, and acceptability of a worksite lifestyle improvement program that includes lifestyle education classes led by trained individuals from the worksite and improvements in the worksite environment that will make it easier for employees at risk for diabetes or with unmedicated diabetes to lose weight, exercise more, and eat a healthier diet. A total of 2000 participants across 10 worksites in South, Central, and East India will be involved in this study.

DETAILED DESCRIPTION:
This study will implement and evaluate in a pre-post design trial the acceptability, delivery, effectiveness, and cost-effectiveness of a worksite-based lifestyle improvement package including a peer-led lifestyle change education program (described below) augmented with changes in the worksite environment that promote social support, healthy eating and exercise. The lifestyle education program will include 2000 adults with prediabetes (HbA1c of 5.7-6.4%) or unmedicated diabetes (HbA1c ≥ 6.5% identified at screening) across ten diverse worksites in India (changes to the worksite environment will impact a much broader population of employees). A mixed methods approach will be used to evaluate implementation of the program.

Participants at high risk for diabetes or with unmedicated diabetes will be enrolled in a lifestyle intervention training program that includes strategies to maintain a healthy weight, maintain healthy blood glucose levels, eat a healthy diet, increase physical activity, overcome barriers, and build social support. Participants will be assigned two goals to achieve during lifestyle classes; to increase the physical activity to at least 150 minutes per week of moderate level activity and lose at least 5% of their baseline body weight. Participants also will be given knowledge and tools necessary to improve their diet quality and quantity.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥23 kg/m2 and/or waist circumference ≥90 cm for men and ≥80 cm for women
* Prediabetic (HbA1c of 5.7-6.4%) or diabetic (HbA1c≥6.5%)

Exclusion Criteria:

* Currently taking any diabetes medications
* Pregnant or breastfeeding
* History of heart disease, current serious illness, or conditions which would impede participation in an unsupervised physical activity and diet change program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2108 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Weber, PhD, Principal Investigator — Emory University
Locations (2):
- India (2):
  - Madras Diabetes Research Foundation, Chennai
  - Public Health Foundation of India, New Delhi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weber MB, Rhodes EC, Ranjani H, Jeemon P, Ali MK, Hennink MM, Anjana RM, Mohan V, Narayan KMV, Prabhakaran D. Adapting and scaling a proven diabetes prevention program across 11 worksites in India: the INDIA-WORKS trial. Implement Sci Commun. 2023 Nov 13;4(1):134. doi: 10.1186/s43058-023-00516-1. PMID 37957783
- [Derived] Weber MB, Rhodes EC, Ranjani H, Jeemon P, Ali MK, Hennink MM, Anjana RM, Mohan V, Narayan KV, Prabhakaran D. Adapting and scaling a proven diabetes prevention program across 11 worksites in India: the INDIA-WORKS trial. Res Sq [Preprint]. 2023 Aug 4:rs.3.rs-3143470. doi: 10.21203/rs.3.rs-3143470/v1. PMID 37577514

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lifestyle Intervention Training Program
Started | 2108
Completed | 1358
Not Completed | 750
Not completed — Death | 4
Not completed — Lost to Follow-up | 509
Not completed — Withdrawal by Subject | 148
Not completed — No longer at worksite | 85
Not completed — Medical reasons not related to the study | 4

BASELINE CHARACTERISTICS:
Arm/Group | Lifestyle Intervention Training Program
Number analyzed (Participants) | 2108
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.83 (8.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 477
  Male | 1631
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2108
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  India | 2108
Number of participants at baseline without known diabetes [Count of Participants; unit: Participants] | 1448

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reaching Two or More Cardiometabolic Risk Goals
Description: The primary outcome assessing program effectiveness is a composite of achieving two or more cardiometabolic risk goals; participants will be scored on the number of risk factors they improve on (0-3) with success delineated by a HbA1c decrease ≥0.5%; a systolic blood pressure decrease ≥5 mm Hg; and a decrease in plasma triglycerides ≥10 mg/dl.
  Number of participants reaching two or more cardiometabolic Risk Goals will be reported.
Time Frame: Annually up to 2 years
Population: Number of participants analyzed in each time point varies from overall number analyzed due to missing samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Intervention Training Program
Number analyzed (Participants) | 1411
Participants
  1 year post-intervention | 485
  2 years post-intervention: number analyzed (Participants) | 1193
  2 years post-intervention | 351

2. Secondary Outcome: Blood Pressure (BP)
Description: Blood pressure in mmHg will be measured with an automated blood pressure machine annually, from baseline to the end of follow-up (up to two years). Blood pressure measurements are as follows:
  Normal = systolic, less than 120 and diastolic, less than 80 Prehypertension = systolic, 120 - 139 or diastolic , 80 - 89 High Blood Pressure/(Hypertension) Stage 1 = systolic, 140 - 159 or diastolic, 90 - 99 High Blood Pressure (Hypertension) Stage 2 = systolic, 160 or higher or diastolic, 100 or higher Hypertensive Crisis (Emergency care needed) = systolic, Higher than 180 or diastolic, Higher than 110
Time Frame: Baseline, Annually up to 2 years
Population: Number of participants analyzed in each row differ from overall number analyzed due to patients unable to complete the visit or unable to provide the BP measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lifestyle Intervention Training Program
Number analyzed (Participants) | 2108
mmHg
  Baseline Systolic Blood Pressure | 132.28 (16.64)
  Systolic Blood Pressure at 1 year post-intervention: number analyzed (Participants) | 1379
  Systolic Blood Pressure at 1 year post-intervention | 127 (14.28)
  Systolic Blood Pressure at 2 years post-intervention: number analyzed (Participants) | 1143
  Systolic Blood Pressure at 2 years post-intervention | 128.4 (15.0)
  Baseline Diastolic Blood Pressure | 85.21 (10.36)
  Diastolic Blood Pressure at 1 year post-intervention: number analyzed (Participants) | 1379
  Diastolic Blood Pressure at 1 year post-intervention | 83.6 (9.4)
  Diastolic Blood Pressure at 2 years post-intervention: number analyzed (Participants) | 1143
  Diastolic Blood Pressure at 2 years post-intervention | 83.8 (9.50)

3. Secondary Outcome: Mean Hemoglobin A1c (HbA1c) Level
Description: HbA1c will be assessed via blood draw and processing annually, from baseline to the end of study follow-up (up to 2 years).
Time Frame: Baseline, annually up to 2 years
Population: Number analyzed in one or more rows differs from overall number analyzed due to lost to follow up patients and missing samples.
Measure: Mean (Standard Deviation); unit: percentage of HbA1C
Arm/Group | Lifestyle Intervention Training Program
Number analyzed (Participants) | 2108
percentage of HbA1C
  Baseline HbA1c (%) | 6.41 (0.97)
  Ave HbA1c (%) at 1 year follow-up visit: number analyzed (Participants) | 1418
  Ave HbA1c (%) at 1 year follow-up visit | 6.1 (1.1)
  Ave HbA1c (%) at 2 years follow-up: number analyzed (Participants) | 1284
  Ave HbA1c (%) at 2 years follow-up | 6.3 (1.2)

4. Secondary Outcome: Number of New Diabetes Cases
Description: Number of new cases of diabetes is the number of participants diagnosed with a new onset of diabetes using the HbA1c test (HbA1c levels of 6.5% or higher indicate diabetes). Number of new cases of diabetes will be collected annually, from baseline to the end of study follow-up (up to 2 years).
Time Frame: Baseline, end of follow up (up to 2 years post-baseline)
Population: Number analyzed at ave 2 years post-intervention included number of participants that completed the ave 2 years post-intervention visit and provided data for diabetes incidence.
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Intervention Training Program
Number analyzed (Participants) | 2108
Participants
  Baseline | 660
  End of study follow-up (up to 2 years post-baseline): number analyzed (Participants) | 1448
  End of study follow-up (up to 2 years post-baseline) | 481

5. Secondary Outcome: Mean Fasting Plasma Glucose
Description: Fasting plasma glucose will be assessed via blood draw. Fasting plasma glucose will be collected annually, from baseline to the end of study follow-up (up to 2 years). A normal fasting blood sugar on awakening is less under 100 mg/dl.
Time Frame: Baseline, annually up to 2 years
Population: Number analyzed in one or more rows differs from overall number analyzed due to missing blood samples for this outcome and patients that were lost to follow up.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Lifestyle Intervention Training Program
Number analyzed (Participants) | 2108
mg/dl
  Baseline Mean Fasting Plasma Glucose: number analyzed (Participants) | 1628
  Baseline Mean Fasting Plasma Glucose | 105.80 (27.75)
  Mean Fasting Plasma Glucose at Ave 1 year post-intervention: number analyzed (Participants) | 1356
  Mean Fasting Plasma Glucose at Ave 1 year post-intervention | 108.6 (33.6)
  Mean Fasting Plasma Glucose at Ave 2 years post-intervention: number analyzed (Participants) | 1030
  Mean Fasting Plasma Glucose at Ave 2 years post-intervention | 113.6 (37.5)

6. Secondary Outcome: Mean Body Mass Index (BMI)
Description: BMI will be calculated in kg/m^2 from annual measures of height (m) and weight (kg). BMI will be collected annually, from baseline to the end of study follow-up (up to 2 years).
Time Frame: Baseline, Annually up to 2 years
Population: Number analyzed in one or more rows differs from overall number analyzed due to patients unable to complete the study visit and provide data for this outcome.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Lifestyle Intervention Training Program
Number analyzed (Participants) | 2108
kg/m^2
  Baseline | 27.35 (3.61)
  1 year post-intervention: number analyzed (Participants) | 1378
  1 year post-intervention | 27.2 (3.7)
  2 years post-intervention: number analyzed (Participants) | 1238
  2 years post-intervention | 27.1 (3.7)

7. Secondary Outcome: Mean Body Weight
Description: Weight will be measured in kilograms using a digital scale. Weight will be collected annually post-intervention from baseline to the end of study follow-up (up to 2 years).
Time Frame: Baseline, Annually up to 2 years
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Lifestyle Intervention Training Program
Number analyzed (Participants) | 2108
Kg
  Baseline body weight | 74.2 (12.4)
  1 year post-intervention: number analyzed (Participants) | 1381
  1 year post-intervention | 73.4 (12.5)
  2 years post-intervention: number analyzed (Participants) | 1255
  2 years post-intervention | 72.7 (12.2)

8. Secondary Outcome: Waist Circumference
Description: Waist circumference will be measured in centimeters using a non-elastic measuring tape. Waist circumference will be collected annually, from baseline to the end of study follow-up (up to 2 years).
Time Frame: Baseline, Annually up to 2 years
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Lifestyle Intervention Training Program
Number analyzed (Participants) | 2108
cm
  Baseline | 95.5 (8.9)
  1 year post-intervention: number analyzed (Participants) | 1377
  1 year post-intervention | 93.7 (9.1)
  2 years post-intervention: number analyzed (Participants) | 1137
  2 years post-intervention | 94.0 (9.2)

9. Secondary Outcome: Number of Patients Overweight or Obese
Description: The number of participants of participants who are overweight or obese will be calculated from the body mass index annually, from baseline to the end of study follow-up (up to two years). Overweight and Obesity will be defined using WHO-recommended outpoints for Asian populations: overweight = BMI of 23-<27.5 kg/m^2 and obese = BMI of 27.5 kg/m2 or greater.
Time Frame: Baseline, Annually up to 2 years
Population: Number analyzed in each time point include patients that completed each follow up visit and where able to provide data about the weight.
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Intervention Training Program
Number analyzed (Participants) | 2108
Participants
  Overweight patients at Baseline | 639
  Overweight patients at 1 year post-intervention: number analyzed (Participants) | 1378
  Overweight patients at 1 year post-intervention | 653
  Overweight patients at 2 years post-intervention: number analyzed (Participants) | 1238
  Overweight patients at 2 years post-intervention | 604
  Obese patients at Baseline | 863
  Obese patients at 1 year post-intervention: number analyzed (Participants) | 1378
  Obese patients at 1 year post-intervention | 604
  Obese patients at 2 years post-intervention: number analyzed (Participants) | 1238
  Obese patients at 2 years post-intervention | 524

10. Secondary Outcome: Prevalence of Hypertension
Description: Number of participants with hypertension will be calculated from annual blood pressure measurements, from baseline to the end of study follow-up (up to two years). Hypertension is defined as the following: Stage 1: systolic 140 - 159 mmHg or diastolic 90 - 99 mmHg; Stage 2: systolic 160 mmHg or higher, or diastolic 100 mmHg or higher; hypertensive crisis (emergency care needed): systolic higher than 180 mmHg or diastolic higher than 110 mmHg.
Time Frame: Annually up to 2 years
Population: Number analyzed in each time point include patients that completed each follow up visit and where able to provide data about Blood Pressure.
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Intervention Training Program
Number analyzed (Participants) | 1379
Participants
  Any Hypertension at 1 year post-intervention | 388
  Hypertension Stage 1 at 1 year post-intervention | 307
  Hypertension Stage 2 at 1 year post-intervention | 68
  Hypertension Crisis at 1 year post-intervention | 13
  Any Hypertension at 2 years post-intervention: number analyzed (Participants) | 1143
  Any Hypertension at 2 years post-intervention | 357
  Hypertension Stage 1 at 2 years post-intervention: number analyzed (Participants) | 1143
  Hypertension Stage 1 at 2 years post-intervention | 280
  Hypertension Stage 2 at 2 years post-intervention: number analyzed (Participants) | 1143
  Hypertension Stage 2 at 2 years post-intervention | 64
  Hypertension Crisis at 2 years post-intervention: number analyzed (Participants) | 1143
  Hypertension Crisis at 2 years post-intervention | 13

11. Secondary Outcome: Mean Triglycerides Level
Description: Plasma triglycerides will be assessed via blood draw and will be assessed annually, from baseline to the end of study follow-up (up to two years).
Time Frame: Baseline, annually up to 2 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Lifestyle Intervention Training Program
Number analyzed (Participants) | 2108
mg/dl
  Baseline: number analyzed (Participants) | 1630
  Baseline | 140.58 (85.53)
  1 year post-intervention: number analyzed (Participants) | 1398
  1 year post-intervention | 148.8 (95.2)
  2 years post-intervention: number analyzed (Participants) | 1189
  2 years post-intervention | 155.8 (89.0)

12. Secondary Outcome: Mean Low Density Lipoprotein (LDL)
Description: LDL cholesterol will be assessed via blood draw and will be measured annually, from baseline to the end of study follow-up (up to two years).
Time Frame: Baseline, Annually up to 2 years
Population: Number analyzed in one or more rows differs from overall number analyzed due to missing samples and lost to follow up patients.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Lifestyle Intervention Training Program
Number analyzed (Participants) | 1630
mg/dl
  Baseline LDL | 117.0 (35.3)
  1 year post-intervention: number analyzed (Participants) | 1398
  1 year post-intervention | 119.0 (35.8)
  2 years post-intervention: number analyzed (Participants) | 1183
  2 years post-intervention | 121.6 (34.7)

13. Secondary Outcome: Mean High Density Lipoprotein (HDL)
Description: HDL cholesterol will be assessed via blood draw and will be measured annually, from baseline to the end of study follow-up (up to 2 years).
Time Frame: Baseline, Annually up to 2 years
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Lifestyle Intervention Training Program
Number analyzed (Participants) | 1630
mg/dl
  Baseline | 43.54 (9.18)
  1 year-post-intervention: number analyzed (Participants) | 1398
  1 year-post-intervention | 44.2 (9.2)
  2 years post-intervention: number analyzed (Participants) | 1189
  2 years post-intervention | 43.9 (9.7)

14. Secondary Outcome: Number of Patients With Prediabetes or Newly Detected Diabetes That Achieve Normoglycemia Rates
Description: Number of participants with Dysglycemia (HbA1c > 5.7%) that reach normoglycemia (HbA1c < 5.7%) at the end of the study (up to two years).
Time Frame: End of study follow-up (Up to 2 years post-intervention)
Population: The overall number of participants analyzed in this outcome refers to the number of patients at baseline without known diabetes.
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Intervention Training Program
Number analyzed (Participants) | 1448
Participants | 330

ADVERSE EVENTS:
Time Frame: 2 years post-intervention
Arm/Group | Lifestyle Intervention Training Program
All-Cause Mortality (participants affected / at risk) | 4/2108
Serious Adverse Events (participants affected / at risk) | 0/2108
Other Adverse Events (participants affected / at risk) | 0/2108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/68/NCT02813668/Prot_SAP_001.pdf
  • Informed Consent Form (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT02813668/ICF_000.pdf